CLINICAL TRIAL: NCT04844138
Title: Evaluating a Self-Directed Cognitive Behavioural Therapy E-Health and M-Health Program for Anxiety in Pregnancy and Postpartum During COVID-19
Brief Title: Evaluating Overcoming Anxiety in Pregnancy and Postpartum as an Online Self-Directed Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Kristin Reynolds, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P2020:104; 53294 (Other Grant/Funding Number: Research Manitoba)
Record Dates: First submitted 2021-04-05; First posted 2021-04-14 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Perinatal Anxiety; Perinatal Depression
Keywords: Anxiety; Pregnancy; Postpartum; Online; Self-Directed; Cognitive Behavioural Therapy; Randomized Controlled Trial; COVID-19
MeSH Terms: conditions — Anxiety Disorders; COVID-19 | interventions — Pregnancy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the online self-directed program condition or the waitlist condition. Throughout the study, participant outcomes for both conditions will be measured to evaluate the effects of our online program compared to treatment as usual.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The research team (principal investigator, co-investigators, research coordinator, and research assistants) will be blinded during the randomization process. To protect participants' identifying information throughout the study, a non-team member will generate a randomized list of unique participant IDs prior to starting recruitment. The non-team member will then randomly assign these IDs to the online self-directed program or waitlist conditions, and will black out this information to conceal it from the research team. The research coordinator will assign participants to a participant ID when they are enrolled in our study. After participants complete their second screening interview (clinical symptom interview), the research coordinator will access the blacked-out information and reveal the participant's condition. Once revealed, this information may be viewed by all members of the research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Self-Directed Program (Experimental): Participants in this condition will complete our six-week online self-directed program as soon as it's available.
  Interventions: Behavioral: Overcoming Anxiety in Pregnancy and Postpartum Online Self-Directed Program
- Waitlist (Other): Participants in this condition will receive treatment as usual for six weeks, after which point they will be invited to complete our online program.
  Interventions: Behavioral: Overcoming Anxiety in Pregnancy and Postpartum Online Self-Directed Program

INTERVENTIONS:
Behavioral: Overcoming Anxiety in Pregnancy and Postpartum Online Self-Directed Program — The investigators will administer the Overcoming Anxiety in Pregnancy and Postpartum program in an online self-directed format. This program is grounded in Cognitive Behavioural Therapy and will teach participants strategies to manage their anxiety. Participants will complete six modules that will be released to them on a bi-weekly basis.

SUMMARY:
The pregnancy and postpartum periods can be joyous times in life; however, they can also be filled with challenging physical, emotional, and lifestyle changes. These changes may lead to feelings of stress, anxiety, and depression amongst new and expecting mothers, which can have negative effects on fetal and infant development (Beijers et al., 2010; Goodman et al., 2016). The impacts of increased worry about health and safety due to COVID-19 as well as future-related uncertainties, paired with social (physical) distancing, may be felt especially strongly in this population. Of concern, pregnant and postpartum women have low rates of mental health service use even prior to the pandemic (Fonseca et al., 2015). E-health (Internet) and m-health (mobile application) psychological interventions are accessible, available at reduced cost, and can be accessed within users' homes, a factor that is particularly important during the pandemic (Andrews & Titov, 2010). In this study, the investigators will disseminate a free, online, self-directed Cognitive Behavioural Therapy program to women experiencing symptoms of anxiety during pregnancy and postpartum. This program has shown to be effective at improving symptoms of anxiety and depression when delivered in an in-person group format, and has high acceptability (Furer & Reynolds, 2015). The investigators will transfer this program into an online format so that pregnant and postpartum users can navigate the sessions on their own, without the support of a clinician. This program contains six modules which include topics such as coping with negative thoughts, unpacking the myth of the supermom, and managing expectations during pregnancy and postpartum. Additionally, material related to COVID-19 has been added to the program to target any pandemic-related stress participants may be experiencing. The investigators will collect information about the program's feasibility, acceptability, and effectiveness, which will inform future improvements to the program. This program is expected to reduce participants' feelings of stress, anxiety, and depression, in addition to improving maternal attachment. It is anticipated that these gains will be maintained when the investigators follow-up with participants one month after program completion. This program has the potential to provide accessible and affordable mental health services to pregnant and postpartum women struggling during the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant or within 12 months postpartum
* Age 18 or older
* Experiencing symptoms of anxiety
* Have access to a computer, tablet, or smartphone
* Have access to the Internet
* Speak English
* Manitoba resident
* Willing to provide their name, email address, home address, and phone number

Exclusion Criteria:

* Current substance use disorder
* Diagnoses of bipolar disorder or schizophrenia
* Current suicidality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Change in Perinatal Anxiety Symptoms from Baseline | The online self-directed program condition will complete it at weeks 1, 6, and 10, while the waitlist condition will complete it at weeks 1, 6, 12, and 16. Both conditions will complete the short version weekly during the program.
  To assess changes in perinatal anxiety symptoms throughout the study, the Perinatal Anxiety Screening Scale (PASS; Somerville et al., 2014) will be administered. The PASS is a 31-item self-report measure assessing symptoms of anxiety during the perinatal period. The scale has excellent reliability, adequate test-retest reliability, and strong evidence of convergent validity (Somerville et al., 2014). A shortened version of the PASS will be administered to participants in both conditions when they are completing the online program. This measure will help determine the effectiveness of this program.

SECONDARY OUTCOMES:
Change in Perinatal Depression Symptoms from Baseline | The online self-directed program condition will complete it at weeks 1, 6, and 10, while the waitlist condition will complete it at weeks 1, 6, 12, and 16. Both conditions will complete it weekly during the program.
  To examine changes in perinatal depression symptoms throughout the study, the Edinburgh Postnatal Depression Scale (Cox et al., 1987) will be administered. The EPDS is a 10-item self-report measure assessing symptoms of postnatal depression on a 0 to 4 scale. Higher scores indicate higher levels of depression symptoms. This scale exhibits satisfactory psychometric properties and is sensitive to change (Cox et al., 1987). It has also been validated in pregnant populations. The investigators have removed item 10 (suicidality measure) as participants with suicidal ideations will be screened out at the initial screening interview. This outcome measure will help determine the effectiveness of this program.
Change in COVID-19 Stress from Baseline | The online self-directed program condition will complete it at weeks 1, 6, 10, while the waitlist condition will complete it at weeks 1, 6, 12, and 16.
  To assess changes in COVID-19 related stress, the COVID-19 Stress Scales (Taylor et al., 2020) will be administered. This is a 36-item measure, with higher scores indicating higher levels of stress. It measures specific factors that may contribute to pandemic-related distress, including danger and contamination fears, fears about the socio-economic consequences of the pandemic, xenophobia (i.e. foreigners carrying the disease), compulsive checking and reassurance seeking, and traumatic stress symptoms about the virus. When tested in a North American sample, these scales were found to be intercorrelated and had acceptable reliability and validity (Taylor et al., 2020). This outcome measure will help determine the effectiveness of this program.
Change in Non-Specific Psychological Distress from Baseline | The online self-directed program condition will complete it at weeks 1, 6, 10, while the waitlist condition will complete it at weeks 1, 6, 12 and 16.
  To assess changes in non-specific psychological distress across this study, the Kessler Distress Scale-Short Form-6-item version (K6; Kessler et al., 2002) will be administered. The K6 is a 6-item self-report measure and has been shown to have excellent internal reliability. This outcome measure will help determine the effectiveness of this program.
Change in Life Stress from Baseline | The online self-directed program condition will complete it at weeks 1, 6, 10, while the waitlist condition will complete it at weeks 1, 6, 12, and 16.
  To assess changes in life stress across this study, the Perceived Stress Scale (PSS; Cohen et al., 1983) will be administered. The PSS is a 10-item self-report measure that assesses the extent to which one's life is appraised as stressful. This outcome measure will help determine the effectiveness of this program.
Change in Maternal Antenatal Attachment from Baseline | The online self-directed program condition will complete it at weeks 1, 6, 10, while the waitlist condition will complete it at weeks 1, 6, 12, and 16.
  To evaluate changes in maternal antenatal attachment throughout this study, the Maternal Antenatal Attachment Scale (MAAS; Condon, 1993) will be administered to pregnant participants in both conditions. The MAAS is a 15-item self-report measure that assesses maternal attachment towards an unborn baby in the antenatal period. This outcome measure will help determine the effectiveness of this program.
Change in Maternal Postnatal Attachment from Baseline | The online self-directed program condition will complete it at weeks 1, 6, 10, while the waitlist condition will complete it at weeks 1, 6, 12, and 16.
  To evaluate changes in maternal antenatal attachment throughout this study, the Maternal Antenatal Postnatal Scale (MPAS; Condon & Corkindale, 1998) will be administered to postpartum participants in both conditions. The MPAS is a 19-tem self-report measure that assesses maternal attachment towards an infant during the postnatal period. This outcome measure will help determine the effectiveness of this program.
Change in Maternal Efficacy from Baseline | The online self-directed program condition will complete it at weeks 1, 6, 10, while the waitlist condition will complete it at weeks 1, 6, 12, and 16.
  To evaluate changes in maternal efficacy throughout this study, the Maternal Efficacy Questionnaire (MEQ; Teti & Gelfand, 1991) will be administered to postpartum participants in both conditions. The MEQ is a 10-item self-report measure that assesses a mother's perception of her own parenting competence. This outcome measure will help determine the effectiveness of this program.
Acceptability of the Online Self-Directed Program | The TAAS will be administered to the online self-directed program condition at week 2 and the waitlist condition at week 7.
  To assess the acceptability of our online self-directed program, the Treatment Acceptability/Adherence Scale (TAAS; Milosevic et al., 2015) will be administered. The TAAS is a self-report measure of treatment acceptability which exhibits sound psychometric properties. The TAAS will be administered to participants in both conditions once they have completed the second module of the online program. This measure will help determine the acceptability of this program with pregnant and postpartum persons.
Participant Satisfaction with the Online Self-Directed Program | This measure will be administered to the online self-directed program condition at program completion (week 6) and to the waitlist condition at program completion (week 12).
  To assess participants' satisfaction with the Overcoming Anxiety in Pregnancy and Postpartum online self-directed program, the Treatment Satisfaction Measure (Furer & Reynolds, 2015) will be administered. This measure was created for the Overcoming Anxiety in Pregnancy and Postpartum Group Treatment Program and has been adapted for this online program. Two items ask about the helpfulness of the workbook and its focus on perinatal issues and are rated on a 5-point scale (i.e., from "very helpful" to "not at all helpful"). Two additional yes/no questions are included, regarding whether participants would recommend the program to other individuals in the perinatal period and whether they themselves would participate in the program again if needed. Two final open-ended questions are included regarding what patients liked about the program, and any suggestions they would have for changes to it.
Participant Experiences in the Online Self-Directed Program | The weekly feedback measure will be administered weekly during the program (online self-directed program condition: weeks 1-6; waitlist condition: weeks 6-12). The interview will take place at week 6.
  To obtain more detailed feedback from participants about their experiences in this online program, the investigators have developed a weekly feedback measure. This measure asks participants about their engagement with each module and allows them to provide specific feedback about the content of each module. The investigators will also invite 25 participants from each condition to complete a qualitative interview to discuss their experiences in the program and on the waitlist for the program. This will allow the investigators to collect more detailed data about what participants (dis)liked about the online program. This data will allow the investigators to improve the program for future users.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Reynolds, Ph.D., Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrews G, Titov N. Is internet treatment for depressive and anxiety disorders ready for prime time? Med J Aust. 2010 Jun 7;192(S11):S45-7. doi: 10.5694/j.1326-5377.2010.tb03693.x. PMID 20528709
- [Background] Beijers R, Jansen J, Riksen-Walraven M, de Weerth C. Maternal prenatal anxiety and stress predict infant illnesses and health complaints. Pediatrics. 2010 Aug;126(2):e401-9. doi: 10.1542/peds.2009-3226. Epub 2010 Jul 19. PMID 20643724
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Condon JT. The assessment of antenatal emotional attachment: development of a questionnaire instrument. Br J Med Psychol. 1993 Jun;66(2):167-83. doi: 10.1111/j.2044-8341.1993.tb01739.x. PMID 8353110
- [Background] Condon JT, Corkindale CJ. The assessment of parent-to-infant attachment: Development of a self-report questionnaire instrument. Journal of Reproductive and Infant Psychology. 1998; 16(1): 57-76.
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Fairbrother N, Janssen P, Antony MM, Tucker E, Young AH. Perinatal anxiety disorder prevalence and incidence. J Affect Disord. 2016 Aug;200:148-55. doi: 10.1016/j.jad.2015.12.082. Epub 2016 Apr 14. PMID 27131505
- [Background] Fonseca A, Gorayeb R, Canavarro MC. Women׳s help-seeking behaviours for depressive symptoms during the perinatal period: Socio-demographic and clinical correlates and perceived barriers to seeking professional help. Midwifery. 2015 Dec;31(12):1177-85. doi: 10.1016/j.midw.2015.09.002. Epub 2015 Sep 21. PMID 26433622
- [Background] Furer P, Reynolds K. Overcoming anxiety in pregnancy and postpartum. Unpublished treatment manual. Winnipeg, MB: University of Manitoba; 2015.
- [Background] Gavin NI, Gaynes BN, Lohr KN, Meltzer-Brody S, Gartlehner G, Swinson T. Perinatal depression: a systematic review of prevalence and incidence. Obstet Gynecol. 2005 Nov;106(5 Pt 1):1071-83. doi: 10.1097/01.AOG.0000183597.31630.db. PMID 16260528
- [Background] Goodman JH, Watson GR, Stubbs B. Anxiety disorders in postpartum women: A systematic review and meta-analysis. J Affect Disord. 2016 Oct;203:292-331. doi: 10.1016/j.jad.2016.05.033. Epub 2016 Jun 1. PMID 27317922
- [Background] Kessler RC, Andrews G, Colpe LJ, Hiripi E, Mroczek DK, Normand SL, Walters EE, Zaslavsky AM. Short screening scales to monitor population prevalences and trends in non-specific psychological distress. Psychol Med. 2002 Aug;32(6):959-76. doi: 10.1017/s0033291702006074. PMID 12214795
- [Background] Milosevic I, Levy HC, Alcolado GM, Radomsky AS. The Treatment Acceptability/Adherence Scale: Moving Beyond the Assessment of Treatment Effectiveness. Cogn Behav Ther. 2015;44(6):456-69. doi: 10.1080/16506073.2015.1053407. Epub 2015 Jun 19. PMID 26091250
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Somerville S, Dedman K, Hagan R, Oxnam E, Wettinger M, Byrne S, Coo S, Doherty D, Page AC. The Perinatal Anxiety Screening Scale: development and preliminary validation. Arch Womens Ment Health. 2014 Oct;17(5):443-54. doi: 10.1007/s00737-014-0425-8. Epub 2014 Apr 4. PMID 24699796
- [Background] Taylor S, Landry CA, Paluszek MM, Fergus TA, McKay D, Asmundson GJG. Development and initial validation of the COVID Stress Scales. J Anxiety Disord. 2020 May;72:102232. doi: 10.1016/j.janxdis.2020.102232. Epub 2020 May 4. PMID 32408047
- [Background] Teti DM, Gelfand DM. Behavioral competence among mothers of infants in the first year: the mediational role of maternal self-efficacy. Child Dev. 1991 Oct;62(5):918-29. doi: 10.1111/j.1467-8624.1991.tb01580.x. PMID 1756667
- [Derived] Uchechukwu L, Hardman MP, Hadley I, Gornik ME, Petty SK, Pryor TAM, Alcolado GM, Furer P, Reynolds KA. "I'm not alone": perinatal women's experiences in an online self-directed program for perinatal anxiety. BMC Pregnancy Childbirth. 2025 Feb 21;25(1):190. doi: 10.1186/s12884-025-07270-3. PMID 39984893